CLINICAL TRIAL: NCT06627621
Title: EVALUATION of the EFFICACY of E-POLYCAPROLACTONE-CONTAINING MEMBRANE in ALVEOLAR BONE REGENERATION: a RETROSPECTIVE STUDY
Brief Title: E-Polycaprolactone-Containing Membrane in Alveolar Bone Regeneration
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: cem üngör (Other)
Responsible Party: Sponsor-Investigator, cem üngör, Professor Dr Cem UNGOR, Karadeniz Technical University
Organization: Karadeniz Technical University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023/20
Record Dates: First submitted 2024-10-03; First posted 2024-10-04 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Alveolar Bone Grafting
Keywords: alveolar ridge augmentation, alveolar bone loss, dental implant, guided tissue regeneration, polycaprolactone
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (1):
- Alveolar bone grafting (Other): Scaffold guided bone regeneration
  Interventions: Procedure: Alveolar Ridge Reconstruction

INTERVENTIONS:
Procedure: Alveolar Ridge Reconstruction — scaffold guided alveolar bone regeneration

SUMMARY:
This study aimed to evaluate the effectiveness of synthetic polycaprolactone (PCL) bioscaffold membranes used for alveolar augmentation in maxillofacial surgery for increasing the amount of newly formed bone after three-dimensional application.

ELIGIBILITY:
Inclusion Criteria:

* (1) patients aged >18 years without any systemic disease or with an established systemic disease that precluded the surgical procedure; (2) patients whose bone deficiency was augmented with PCL scaffolds; (3) patients with an indication for dental implant-supported prosthesis who lacked sufficient bone for dental implants according to cone beam computed tomography (CBCT) evaluation and, therefore, needed bone augmentation; and (4) patients with preoperative and postoperative images.

Exclusion Criteria:

* patients (1) with uncontrolled systemic diseases, (2) who had undergone radiation therapy, (3) who were female and pregnant, (4) who had previously undergone any surgical procedure related to augmentation in the area of the defect, (5) who had incomplete files or lacked pre- and post-treatment radiologic records, or (6) who had psychological problems.

Ages: 18 Months to 80 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 4 (Actual)
Dates: Start 2021-03-08 (Actual); Primary Completion 2023-01-08 (Actual); Study Completion 2023-01-08 (Actual)

PRIMARY OUTCOMES:
Shapiro-Wilk test | From enrollment to the end of treatment at 6 months
  Descriptive statistics are presented as median, mean, standard deviation, minimum-maximum, standard error, and frequency values

CONTACTS AND LOCATIONS:
Locations (1):
- Karadeniz Technical University, Faculty of Dentistry, Department of Oral and Maxillofacial Surgery, Trabzon, Trabzon, Turkey (Türkiye)